CLINICAL TRIAL: NCT04194164
Title: Fluid Intake App for Management of Volume Intake in Patients Receiving Chronic Hemodialysis Therapy, Full Scale Trial
Brief Title: Development of Fluid Intake App for Management of Fluid Intake During Hemodialysis , Full Scale Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00048561a
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-09

CONDITIONS: Weight Gain
Keywords: Hemodialysis; End stage renal disease on dialysis; Fluid intake; Interdialytic weight gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: Comparison of interdialytic weight gain with fluid intake as recorded by fluid app
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid intake app (Experimental): Participants in this arm will use the fluid intake app to help them decrease interdialytic fluid intake. Participants will take a survey to assess the efficacy of the fluid app..
  Interventions: Other: Fluid intake app

INTERVENTIONS:
Other: Fluid intake app — Monitor fluid intake and interdialytic weight gain in patients using the fluid app

SUMMARY:
Methods are needed to help decrease interdialytic weight gains in hemodialysis patients. One potential method for accomplishing this goal is to develop an app for smartphones that allow patients to track their fluid intake throughout the course of the day. NCT 03759847 was designed to test the safety and efficacy of this app. In this protocol, part of the same IRB number, patients with large interdialytic fluid gains (3.5% or greater) will use the app to to determine the association between the interdialytic weight gain and the fluid consumed as recorded by use of the app for each interdialytic period.

DETAILED DESCRIPTION:
In this full scale study, the app will be used to try and influence fluid intake behavior in those patients who are identified to have large fluid weight gains, as defined by a greater than 4% increase in interdialytic weight.

There will be two parts to the full scale trial. In the first part of the full scale study, denoted as the active phase, which will last for two months, study participants will be encouraged to use the app on a daily basis and will meet with the study coordinator on weeks 1, 2, 4, 6, and 8 to further assist the participant in decreasing fluid intake between dialysis sessions. In the second portion of the study, denoted as the passive phase, which will last for six months, the patient will use the app and meet with the study coordinator only when requested by the patient. The number of these sessions will be recorded. At the end of the six month passive phase, the participant will meet for the last time with the study coordinator. During each study visit, subjects will be asked to transfer the data from the App to the study coordinator via the data export function of the app.

ELIGIBILITY:
Inclusion Criteria:

* Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective and having given written (dated and signed) informed consent form to take part in the study.
* Adult chronic hemodialysis patient who is at least 18 years of age
* Average interdialytic fluid gains of 3.5% or greater of body weight for both weekdays and weekends for a 30 day period
* Availability of interdialytic weight gains for the 2 month period prior to enrollment into the study
* Access to a smartphone for use of the app and comfort with using apps on a regular basis
* Access to a smartphone running under either iOS or Android operating systems
* Sufficient knowledge and understanding of the English language to use the application available only in English (US) language
* Mental capacity to use and understand the fluid management app
* Willingness to share intake data collected with the research team

Exclusion Criteria:

* Scheduled for a living related renal transplant in the next seven months
* Hospitalization within 30 days of entry into the study
* Current participation in a randomized clinical trial or in the exclusion period of another clinical trial
* Vulnerable subjects defined as individuals whose willingness to volunteer in the clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Mean intradialytic weight gain | between baseline (pre-app) and the Active phase (months 1 and 2)
  Comparison of interdialytic weight change before and during use of the app
Mean intradialytic weight gain | between baseline (pre-app) and the Passive phase (month 3-8)
  Comparison of interdialytic weight change before and during use of the app

SECONDARY OUTCOMES:
Mean intradialytic weight gain | between baseline (pre-app) and the Active phase (months 1 and 2), between baseline (pre-app) and the Passive phase (month 3-8)
25th percentile of intradialytic weight gain | between baseline (pre-app) and the Active phase (months 1 and 2), between baseline (pre-app) and the Passive phase (month 3-8)
75th percentile of intradialytic weight gain | between baseline (pre-app) and the Active phase (months 1 and 2), between baseline (pre-app) and the Passive phase (month 3-8)
Number of days of app usage | the Active phase (months 1 and 2), Passive phase (month 3 through month 8)
Percentage of days of app usage | the Active phase (months 1 and 2), Passive phase (month 3 through month 8)
Number of patients who experienced at least 50% increase in fluid intake during app use | the Active phase (months 1 and 2), Passive phase (month 3 through month 8)
  Safety evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rocco, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Background] 2. United States Renal Data System 2018. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD
- [Background] Eknoyan G, Beck GJ, Cheung AK, Daugirdas JT, Greene T, Kusek JW, Allon M, Bailey J, Delmez JA, Depner TA, Dwyer JT, Levey AS, Levin NW, Milford E, Ornt DB, Rocco MV, Schulman G, Schwab SJ, Teehan BP, Toto R; Hemodialysis (HEMO) Study Group. Effect of dialysis dose and membrane flux in maintenance hemodialysis. N Engl J Med. 2002 Dec 19;347(25):2010-9. doi: 10.1056/NEJMoa021583. PMID 12490682
- [Background] FHN Trial Group; Chertow GM, Levin NW, Beck GJ, Depner TA, Eggers PW, Gassman JJ, Gorodetskaya I, Greene T, James S, Larive B, Lindsay RM, Mehta RL, Miller B, Ornt DB, Rajagopalan S, Rastogi A, Rocco MV, Schiller B, Sergeyeva O, Schulman G, Ting GO, Unruh ML, Star RA, Kliger AS. In-center hemodialysis six times per week versus three times per week. N Engl J Med. 2010 Dec 9;363(24):2287-300. doi: 10.1056/NEJMoa1001593. Epub 2010 Nov 20. PMID 21091062
- [Background] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Schiller BM, Yang PC, Rajagopalan S; Frequent Hemodialysis Network (FHN) Trial Group. Determinants of left ventricular mass in patients on hemodialysis: Frequent Hemodialysis Network (FHN) Trials. Circ Cardiovasc Imaging. 2012 Mar;5(2):251-61. doi: 10.1161/CIRCIMAGING.111.969923. Epub 2012 Feb 23. PMID 22360996
- [Background] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Yang PC, Rajagopalan S; Frequent Hemodialysis Network Trial Group. Effects of frequent hemodialysis on ventricular volumes and left ventricular remodeling. Clin J Am Soc Nephrol. 2013 Dec;8(12):2106-16. doi: 10.2215/CJN.03280313. Epub 2013 Aug 22. PMID 23970131
- [Background] Assimon MM, Wenger JB, Wang L, Flythe JE. Ultrafiltration Rate and Mortality in Maintenance Hemodialysis Patients. Am J Kidney Dis. 2016 Dec;68(6):911-922. doi: 10.1053/j.ajkd.2016.06.020. Epub 2016 Aug 26. PMID 27575009

DOCUMENTS (1):
  • Informed Consent Form (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT04194164/ICF_000.pdf